CLINICAL TRIAL: NCT02388594
Title: A Phase I Study of T-Cells Genetically Modified at the CCR5 Gene by Zinc Finger Nucleases SB-728mR in HIV-Infected Patients, With or Without the CCR5 Delta-32 Mutation, Pre-treated With Cyclophosphamide
Brief Title: A Phase I Study of T-Cells Genetically Modified at the CCR5 Gene by Zinc Finger Nucleases SB-728mR in HIV-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SB-728mR; U01AI104400 (NIH)
Record Dates: First submitted 2015-02-24; First posted 2015-03-17 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Human Immunodeficiency Virus (HIV)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ZFN Modified CD4+ T Cell (Experimental): ZFN Modified CD4+ T Cell
  Interventions: Drug: ZFN Modified CD4+ T Cells
- ZFN Modified CD4+ T Cell with Cyclophosphamide (Experimental): ZFN Modified CD4+ T Cell with Cyclophosphamide
  Interventions: Drug: ZFN Modified CD4+ T Cells; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: ZFN Modified CD4+ T Cells
  Other Names: SB-728mR
Drug: Cyclophosphamide
  Arms: ZFN Modified CD4+ T Cell with Cyclophosphamide

SUMMARY:
This is a triple cohort, open-label pilot study of the safety and antiviral activity of a single infusion of autologous CD4+ T cells genetically modified at the CCR5 gene by Zinc Finger Nucleases SB-728mR (ZFN Modified CD4+ T Cells) using electroporated mRNA with or without the prior administration of two different doses of cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, as documented by a rapid HIV test or any FDA-approved HIV-1 Enzyme or Chemiluminescence Immunoassay (E/CIA) test kit and confirmed by Western blot at any time prior to study entry or HIV antigen, plasma HIV-1 RNA, or second antibody test by a method other than rapid HIV and E/CIA. Alternatively, if a rapid HIV test or any FDA-approved HIV-1 Enzyme or Chemiluminescence Immunoassay (E/CIA) test kit is not available, two HIV-1 RNA values ≥ 2000 copies/mL at least 24 hours apart performed by any laboratory that has CLIA certification, or its equivalent, may be used to document infection.
* CD4+ T cell count of ≥450 cells/mm3 at screen; and a documented CD4 nadir of not lower than 200 cells/mm3.
* Adequate venous access and no other contraindications for leukapheresis.
* Laboratory values obtained at screen:

  1. Hemoglobin: ≥ 10.0 (males); ≥ 9.5 (females) g/dL
  2. Absolute neutrophil count (ANC): ≥ 1000/mm3
  3. Platelet count: ≥ 100,000/mm3
  4. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT): ≤ 2.5 times the upper limit of normal (ULN).
* Subjects must be willing to comply with study-mandated evaluations; including not changing their antiretroviral regimen (unless medically indicated) for 2 months in step 2 or until undergoing the analytical treatment interruption.
* Be male or female, 18 years of age and older.
* Ability and willingness of subject to provide informed consent.
* Have a Karnofsky Performance Score of 70 or higher.
* Have no polymorphisms in the CCR5 ZFN target region as determined by Cel I snp assay at screening.
* Subjects in Cohorts 2 and 3: LVEF > or equal to 40%
* Clinically stable on their first or second HAART regimen. Changes while the patient HIV viral load is undetectable does not count toward the number of ART regimens used, only changes made for virologic failure (for example an individual switching from an NNRTI-based regimen to an integrase inhibitor based regimen while the HIV viral load is undetectable will still be in their first regimen). Site investigator anticipates that a fully active alternative ART regimen could be constructed in the event of virologic failure on the current ART regimen. The current regimen should have no changes within 4 weeks of enrollment. Subjects must be willing to continue on current antiretroviral therapy for the duration of the study except for the duration of the 16 week analytical treatment interruption. NOTE: Subject's ART regimen must be in accordance with the Department of Health and Human Services Document "Guidelines for the Use of Antiretroviral Agents in HIV-1 Infected Adults and Adolescents."
* HIV-1 RNA undetectable by ultrasensitive assay copies/ml obtained at study screening visit or within 60 days prior to study screening visit performed with an ultrasensitive HIV-1 PCR assay. All subjects must have received at least 18 months of therapy and have HIV-1 RNA <50 copies/mL using a FDA-approved assay for at least 48 weeks prior to enrollment. HIV-1 RNA must be measured at least once in the 24 weeks prior to enrollment and at least 3 days before the screening measure. Single determinations that are between ≥50 and <500copies/mL (i.e., blips) are allowed as long as the preceding and subsequent determinations are <50 copies/mL. The screening value may serve as the subsequent determination <50 copies/mL following a blip. NOTE: subjects who have participated in other trials using ATI's will be permitted since detectable virus during the interruption does not represent virologic failure. These subjects should have at least 24 weeks of VL <50 copies/mL.
* Have a recorded viral load set point

Exclusion Criteria:

* Acute or chronic hepatitis B or hepatitis C infection (as further defined in section 6.3.4 and 6.3.8 of this protocol)
* Current or prior AIDS diagnosis.
* History of cancer or malignancy, with the exception of successfully treated basal cell or squamous cell carcinoma of the skin
* History or any features on physical examination indicative of active or unstable cardiac disease or hemodynamic instability. NOTE: subjects with a history of cardiac disease may participate with a physician's approval.
* History or any features on physical examination indicative of a bleeding diathesis.
* Have been previously treated with any HIV experimental vaccine within 6 months prior to screening, or any previous gene therapy using an integrating vector. Note: Subjects treated with placebo in an HIV vaccine study will not be excluded if documentation that they received placebo is provided.
* Use of chronic systemic corticosteroids, hydroxyurea, or immunomodulating agents (e.g., interleukin-2, interferon-alpha or gamma, granulocyte colony stimulating factors, etc.) within 30 days prior to study screening visit. NOTE: Recent or current use of inhaled steroids is not exclusionary. If subjects are prescribed a brief course of oral corticosteroids, the use should be limited to less than 7 days. Use of steroids before apheresis and immune assessment blood draws should be discouraged as it will affect white blood cell function.
* Breast-feeding, pregnant, or unwilling to use acceptable methods of birth control.
* Anticipated use of aspirin, dyprydamole, warfarin or any other medication that is likely to affect platelet function or other aspects of blood coagulation during the 2-week period prior to leukapheresis.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to study screening visit.
* Asymptomatic baseline serum chemistry elevations in LFTs, bilirubin, lipase and serum creatinine due to HAART medication are not exclusionary, when in the opinion of the investigator, the abnormalities are not attributable to intrinsic hepatorenal disease. Such baseline elevations must be due to HAART.
* Receipt of vaccination within 30 days prior to study screening visit. NOTE: It is recommended that subjects enrolling into this study should have completed their routine vaccinations (hepatitis A, hepatitis B, pneumococcus, and tetanus diphtheria booster) at least 30 days prior to screening for the study.
* Have an allergy or hypersensitivity to study product excipients (human serum albumin, DMSO and Dextran 40).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 6 months post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Tebas P, Jadlowsky JK, Shaw PA, Tian L, Esparza E, Brennan AL, Kim S, Naing SY, Richardson MW, Vogel AN, Maldini CR, Kong H, Liu X, Lacey SF, Bauer AM, Mampe F, Richman LP, Lee G, Ando D, Levine BL, Porter DL, Zhao Y, Siegel DL, Bar KJ, June CH, Riley JL. CCR5-edited CD4+ T cells augment HIV-specific immunity to enable post-rebound control of HIV replication. J Clin Invest. 2021 Apr 1;131(7):e144486. doi: 10.1172/JCI144486. PMID 33571163